CLINICAL TRIAL: NCT06988657
Title: Investigation of Cognitive Functions, Manual Skills and Upper Extremity Muscle Thickness of Geriatric Individuals Living in Nursing Homes and Homes
Brief Title: Upper Extremity and Cognitive Functions in Geriatric Individuals Living in Nursing Homes and at Home
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Busra Seckinogullari Korkusuz, Principal Investigator, Ankara University
Other Study IDs: 604.01.02-419
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Geriatric; Nursing Home Resident

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Community-dwelling older adults
- Nursing Home Residents

SUMMARY:
The aim of this study is to examine the cognitive functions, manual skills and upper extremity muscle thickness of geriatric individuals living in a nursing home and at home. Geriatric individuals with similar demographic characteristics between the ages of 55-80 living in a nursing home and at home will be included in the study. Demographic information of the individuals will be recorded and evaluated. Manual skills of geriatric individuals will be evaluated with Purdue Pegboard Test, hand dynamometer, and pinch meter; cognitive status will be evaluated with STROOP, MoCA tests, and muscle thickness will be evaluated with ultrasound. It is planned to include 100 geriatric individuals in the study. Geriatric family members of Atılım University employees and volunteer geriatric individuals in a nursing home will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 60 and 80 years old
* Score above 21 on the Montreal Cognitive Assessment Scale.

Exclusion Criteria:

* Inability to communicate verbally
* Use of walking aids
* Geriatric individuals with severe visual impairment, neurological disorders and/or congestive heart failure
* Older adults in whom exercise is not recommended.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geriatric individuals living in nursing homes and at home with similar demographic characteristics
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic Evaluation | Baseline
  In this study, ultrasonography (US) will be used to evaluate the upper extremity muscle thickness (forearm, biceps, triceps, deltoid) of the participants.
Purdue Pegboard Test | Baseline
  In this study, the Purdue Pegboard Test will be used to evaluate the fine motor skills and hand-eye coordination of the participants.
Hand Dynamometer | Baseline
  In this study, a dynamometer will be used to evaluate the hand grip strength of the participants.
Pinch Meter | Baseline
  In this study, a pinch meter will be used to assess the finger grip strength of the participants.
Stroop T-Bag Form | Baseline
  In this study, the Stroop Test will be applied to evaluate the cognitive control and attention abilities of the participants.
Montreal Cognitive Assessment | Baseline
  In this study, the Montreal Cognitive Assessment (MoCA) test will be applied to evaluate the general cognitive functions of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Study Chair — Atılım University; Büşra Seçkinoğulları Korkusuz, PhD, Principal Investigator — Ankara University
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mathiowetz V, Kashman N, Volland G, Weber K, Dowe M, Rogers S. Grip and pinch strength: normative data for adults. Arch Phys Med Rehabil. 1985 Feb;66(2):69-74. PMID 3970660
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Result] Gitlin LN, Hauck WW, Dennis MP, Winter L. Maintenance of effects of the home environmental skill-building program for family caregivers and individuals with Alzheimer's disease and related disorders. J Gerontol A Biol Sci Med Sci. 2005 Mar;60(3):368-74. doi: 10.1093/gerona/60.3.368. PMID 15860476